CLINICAL TRIAL: NCT01530152
Title: Method Evaluation Study of Truview PCD Versus MacIntosh Laryngoscope
Brief Title: Method Evaluation Study of Truview Picture Capture Device(PCD) Versus MacIntosh Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Per Henrik Lambert, Senior doctor, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NCT-20110006
Record Dates: First submitted 2012-01-24; First posted 2012-02-09 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Intubation
Keywords: Truwiev PCD laryngoscope; Macintosh laryngoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Truwiev PCD laryngoscope — The aim of the method evaluation study is a comparing study of Truview PCD™ laryngoscope vs. Macintosh laryngoscope. The result of this study will form a basis for a possible recommendation of the Truview PCD™ laryngoscope in our organisation.
  The laryngoscopes are compared according to their ability to visualize the glottis area measured by the Cormack Lehane (CL) grade and the time used to get the best CL grade. (See figure 1.) A registration of any damage of tissue/teeths caused by the laryngoscopes, and a possible decrease of the saturation will also be made.
  Other Names: laryngoscopi; generel anaesthesia; lidocain spray

SUMMARY:
Aim:

The aim of the method evaluation study is a comparing study of Truview PCD™ (Picture Capture Device) laryngoscope vs. Macintosh laryngoscope. The result of this study will form a basis for a possible recommendation of the Truview PCD™ laryngoscope in our organisation.

The laryngoscopes are compared according to their ability to visualize the glottis area measured by the Cormack Lehane (CL) grade and the time used to get the best CL grade.

A registration of any damage of tissue/teeths caused by the laryngoscopes, and a possible decrease of the saturation will also be made.

Hypothesis:

The Truview PCD™ laryngoscope provides a better view of the vocal cords and thereby makes the intubation les difficult.

CL 1 is achieved in 90 percent of intubations with the Macintosh laryngoscope, and the hypothesis of the study is that CL 1 can be increased to 98 percent by use of the Truview PCD™ laryngoscope.

DETAILED DESCRIPTION:
The unexpected difficult intubation is, like the difficult mask ventilation, a feared complication to anaesthesia.

A difficult intubation occurs in approx. 1.2 - 3.8 percent of all anaesthesias .

The standard procedure of intubation in Denmark is to use the curved Macintosh blade. This method, however, has some limits, as it requires a direct view of the area of the vocal cords. For that reason we are looking for new methods of intubation that can give a better overview.

The Truview PCD™ laryngoscope is a commercially available laryngoscope with an integrated optical lens that can be connected to a camera head, and gives a better view of trachea during intubation under a general anaestetic. Furthermore it is possible to connect 8-10 liters of oxygen per minute to the Truview PCD™ laryngoscope, which will prevent fog on the viewtube and slow down the rate of desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age who are to undergo a surgery at the ENT department, Aalborg Hospital.
* Patients who understand and accept the trial information.
* SARI score 2-5.

Exclusion Criteria:

* SARI score 0-1 and > 5.
* A need for acute initiation. (By acute initiation the endotracheal tube will be placed in trachea during the first laryngoscopy without prior spraying with local anesthesia).
* If unexpected difficulties during the initiating anesthesia arise, the trial will be interrupted, and the patient will be treated according to the department's guidelines for the situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cormack Lehane (CL) grade | The seconds during intubation where the anaesthesiologist view the vocal cords to determine the CL grade..
  At the first laryngoscopy the patient is sprayed between plica vocalis with Lidocaine 4%, then the patient is ventilated by a mask. During the next laryngoscopy the intubation is performed (the endotracheal tube is placed in trachea).
  The patients are randomized by lottery as to which laryngoscope to be used first.
  After anesthesia induction, preceded by 3 minutes of preoxygenering, the first laryngoscope is used when spraying the patient with Lidocaine. Subsequently the patient is ventilated for 2 minutes, and then the intubation is performed by using the other laryngoscope.

CONTACTS AND LOCATIONS:
Locations (1):
- Per Henrik Lambert, Aalborg, Ålborg, Denmark